CLINICAL TRIAL: NCT05022862
Title: Economic Incentives and Video Directly Observed Therapy to Promote Adherence to Latent Tuberculosis Infection
Brief Title: Economic Incentives and vDOT for Latent Tuberculosis Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00183013; R01AI162888 (NIH)
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Latent Tuberculosis
Keywords: Video Directly Observed Therapy
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual Care (Active Comparator): Participants will receive routine (non-study directed) medical care for latent tuberculosis infection according to published guidelines, including medication, nurse case management, Tuberculosis health education, and toxicity assessments.
  Interventions: Behavioral: Usual Care
- Video Directly Observed Therapy alone (Active Comparator): Participants in this group will receive the same treatments and education provided to Usual Care Control participants, however treatment will be viewed by video directly observed therapy (video-DOT)
  Interventions: Behavioral: Usual Care; Behavioral: Video Directly Observed Therapy alone
- Video Directly Observed Therapy plus Financial Incentives (Experimental): Participants in this group will receive the same treatments and education provided to Usual Care Control participants, as well as treatment viewed by video DOT. This arm will also earn financial contingent incentives. Participants will receive incentive payments when a submitted video is monitored by a staff member and deemed valid. If a participant fails to submit a video on a medication day or if a submitted video is deemed invalid (i.e., not the correct person or no appropriate ingestion of medication), the participant will not receive the scheduled incentive amount that day and the daily incentive value will be decreased.The participant will have opportunities the next day to again resume adherence. After taking the medication again for one week, participants will earn a reduced incentive until they adhere to the medication schedule for a week.
  Interventions: Behavioral: Usual Care; Behavioral: Video Directly Observed Therapy alone; Behavioral: Video Directly Observed Therapy plus Financial Incentives

INTERVENTIONS:
Behavioral: Usual Care — Medication is dispensed to participant at each visit in 30-60 day supplies by Baltimore City Health Department (BCHD) nurses. For study participants, medication dispensation will occur in medication bottles with MEMS Caps, supplied by the study.
Behavioral: Video Directly Observed Therapy alone — Usual care plus Video-DOT using the emocha platform, a HIPAA compliant commercial platform for video based DOT. The app allows a secure/encrypted video recording to be taken as the participant ingests the medication. Electronic text reminders will be sent to the participant on the smart phone when it is time to take the medication. The participant will record a video of the pill ingestion process. Study staff will verify each video to confirm the video shows the correct person and that the pill was ingested appropriately (according to standardized approach involving visualization of the pills, ingestion and observation of an empty mouth after ingestion).
  Arms: Video Directly Observed Therapy alone; Video Directly Observed Therapy plus Financial Incentives
Behavioral: Video Directly Observed Therapy plus Financial Incentives — Usual care plus video-DOT and financial incentives contingent on adherence verified by video DOT. The amount of the financial incentive that can be earned for future verified doses decreases after a missed dose (video). The amount of the financial incentives increases incrementally back to baseline amount after verification of medication ingestion according to the prescribed schedule for several consecutive doses.
  Arms: Video Directly Observed Therapy plus Financial Incentives

SUMMARY:
The purpose of this study is to evaluate a novel and scalable intervention that combines Video Directly Observed Therapy (vDOT) and financial incentives to promote completion of treatment for latent tuberculosis. Adult participants who are initiating treatment for latent tuberculosis will be recruited from the Baltimore City Health Department. The primary hypothesis is that the incentive intervention will increase the percentage of participants that complete the treatment for latent tuberculosis above the completion rates of participants receiving usual care.

DETAILED DESCRIPTION:
Identifying and treating individuals with latent tuberculosis (TB) (LTBI) is a key strategy to achieve the goal of TB elimination in the US but there are many challenges to achieving this goal. In Baltimore, where this research will be conducted, prior studies suggest 35% of non-US--born individuals may have latent TB. Individuals experiencing homelessness have also been found to be at higher risk for TB infection. However, socioeconomic factors such as poverty, access to care, health literacy, and language or cultural barriers present obstacles to treatment. Treatment for latent TB is rarely a priority for patients with many other competing needs. The length of treatment spans many months, and preliminary data shows that less than half will complete prescribed treatment. To date there are limited interventions shown to be effective in increasing adherence to LTBI therapy. Directly observed therapy (DOT) administered via video (Video-DOT, with case-management) has been shown to be effective at monitoring treatment in active TB, but there is limited data when applied to LTBI. Interventions that provide incentives to patients when they meet required therapeutic goals have been demonstrated extraordinarily effective in promoting therapeutic behavior change in diverse populations.

The goal of this randomized trial is to evaluate two adherence interventions ( Video DOT or Video DOT plus financial incentives) versus Usual Care to promote completion of treatment for latent TB among those found eligible and are prescribed short course therapy (isoniazid+Rifampin(3HR), Isoniazid+rifapentine(3HP), or Rifampin alone(4R)) for LTBI care.

The primary assessment of adherence will be treatment completion which is defined as taking 80% of the prescribed doses of medication, as determined by Medication Event Monitoring System (MEMS) caps (i.e., 10 of 12 doses for participants prescribed weekly doses of rifapentine and isoniazid; 96 of 120 doses for participants prescribed daily doses of rifampin; 67 of 84 doses of daily isoniazid and rifampin

Video directly observed therapy (video-DOT) will use the Electronic Mobile Comprehensive Health Application (emocha) platform. This system provides a HIPAA compliant approach for remote DOT combined with data collection that optimizes TB case management. The Video DOT system is comprised of a smart phone/tablet application used by patients, and a web-based dashboard used by the TB clinic. The patient-side application (app) reminds patients to take their medications on a schedule specified by the clinician. For those randomized to the Video-DOT plus incentives arm, additional financial incentives (provided in real-time) are delivered contingent on verification of medication ingestion by video observation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older,
* diagnosed with latent TB and determined to be appropriate for latent TB treatment by participants clinicians
* reside in Baltimore metro area
* speaks English or Spanish, or a language for which there is a short form available via the Johns Hopkins Medicine Institutional Review Board
* prescribed 3 months Isoniazid/Rifapentine, prescribed 3 months Isoniazid/Rifampin, or 4 months Rifampin

Exclusion Criteria:

* younger than 18 years old
* diagnosed with active TB
* prescribed an alternative treatment regimen for latent TB
* pregnant women (as determined by non-study directed clinical evaluation; BCHD performs urine pregnancy testing on women of child bearing age when indicated)
* participant's spoken language does not have a translated long or short consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Estimated)
Dates: Start 2022-02-07 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Treatment Completion | Up to 6 months
  The primary outcome measure, completion of treatment for latent TB, will be assessed for all participants through MEMS caps. A participant will be considered to have completed treatment for study purposes if he/she takes 80% of the prescribed doses of medication, as determined by MEMS caps (i.e., 10 of 12 doses for participants prescribed weekly doses of rifapentine and isoniazid; 96 of 120 doses for participants prescribed daily doses of rifampin; 67 of 84 doses of daily isoniazid and rifampin

SECONDARY OUTCOMES:
Adherence measurements | Up to 6 months
  We will assess how well adherence measured by video based observation of therapy correspond to MEMS caps data in the Intervention arm
Treatment completion (alternative definition) | Up to 6 months
  We will assess treatment completion using video observed therapy (video verification of ingestion) as an alternative measure of adherence in the intervention arms (i.e. comparing completion between video DOT arm, (80% of prescribed doses taken, and defined by accepted videos] and Usual care [80% of prescribed doses taken measured by MEMS caps])
Costs of the incentive intervention | 5 years
  Assess the costs of the incentive intervention. To estimate the costs of the interventions and standard of care, we will utilize an ingredients approach (i.e. micro-costing) in which costs are determined based on unit prices and quantities used. The costs of administering the different components of video-DOT and the Incentives Interventions, and the Usual Care will be based on a combination of direct observations, project records, and clinic invoices.
Cost-effectiveness of the incentive intervention | 5 years
  We will utilize a decision-analytic model to evaluate and report the cost-effectiveness of the intervention, reported as the incremental cost-effectiveness ratio comparing the interventions to usual care, measured against currently accepted willingness to pay thresholds

CONTACTS AND LOCATIONS:
Overall Officials: Maunank Shah, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Baltimore City Health Department, and Baltimore metropolitan area clinics and health departments, Baltimore, Maryland, United States